CLINICAL TRIAL: NCT03278327
Title: Impact of an Endoscopic Treatment of the Line Z on the Gastronomic Recurrence and the Gastro- Esophageal Reflux Disease in the Care of the Adenocarcinoma of Barrett's Oesophagus
Acronym: B-ARMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-ARMS-IPC 2016-017
Record Dates: First submitted 2017-08-21; First posted 2017-09-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Barrett Esophagus Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic resection (Other)
  Interventions: Procedure: Complete endoscopic resection at Day 1 and months 2, 4, 6 8 and month 10.; Device: Endoscopic resection at month 2 and month 4

INTERVENTIONS:
Procedure: Complete endoscopic resection at Day 1 and months 2, 4, 6 8 and month 10. — Endoscopic resection treatment
Device: Endoscopic resection at month 2 and month 4 — System of endoscopic resection of the mucous hurts which can take several forms according to the technical necessities.
  The device the most used in this case is the system COOK Medical Duett of Laboratories.
  The duration of the treatment will be the same duration as the classic endoscopic resection, that is 30 in 60 minutes.
  The resection will be preceded by injection of physiological salt solution tinged with carmine indigo in the sub-mucous membrane.

SUMMARY:
Barrett's oesophagus is a transformation of the esophageal mucous membrane there intestinal metaplasia under the effect of gastro- esophageal reflux disease (GERD).

This metaplasia can evolve in low grade dysplasia LGD) , high grade dysplasia (HGD) then invasive adenocarcinoma.

The treatment of the HGD of the Barrett is the endoscopic treatment. It is about a superficial treatment of tumor without ganglionar invasion by definition.

The endoscopic treatment of the Barrett began in the 2000s, and showed its long-term efficiency.

The studied factors of recurrences are the length of the Barrett, the influence of the eradication completes of the Barrett besides the eradication of the dysplasia, as well as the duration of spacing of the procedures. An anatomical zone is particularly delicate to treat. It is about the anatomical junction between the oesophagus and the stomach appointed junction oeso-gastric or cardia or line Z.

This almost virtual zone is the site of most of the recurrence. The first cause of the oesophagus of Barrett and of its transformation in HGD is the reflux.

This reflux can be handled by medicinal action inhibitor of the pump with proton (PPI) or by surgery (hemi-fundo plicator). This reflux is probably the cause of the long-term recurrence found in the literature.

The surgery is a good treatment of the reflux with however unsatisfactory long-term results. On the other hand, the surgery is little used after endoscopic treatment of a HGD not to compromise the surveillance and the detection of a second offense potentially masked in the surgical fundo-plicator. The endoscopic treatment of the expensive ebb because of the based necessary material too on a fundo-plicator is complicated with use in reason also of his cost.

The medical treatment by PPI for life, besides his duration and thus the potential hardness for the patient, presents long-term complications recently described.

Effects on the appearance of gastric precancerous lesion is not certain, but this association with an osteoporosis is more proved true.

The PPI could also be a etiologic factor of chronic renal insufficiency and insanity.

An endoscopic treatment describes by Inoue " Anti-Reflux Mucosectomy " ( ARMS) allows to decrease the gastro- esophageal reflux disease.

This treatment is an equivalent of on treatment of the line Z which would at the same time allow to make sure of the decrease of recurrence on the line Z by complete treatment of this one and to handle the reflux of these patients.

In this experimental series, 10 patients having made this endoscopic treatment were able to stop their treatment by PPI.

The purpose of this study will be to make sure of the efficiency of the endoscopic treatment of the reflux by it on treatment of this line Z while decreasing the frequent recurrences on this line Z.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years,
* High grade dysplasia or superficial Barrett's oesophagus adenocarcinoma diagnosis,
* Written informed consent,
* Affiliation to Social Security System.

Exclusion Criteria:

* Hiatal hernia,
* Surgical histories treatment of gastro- esophageal reflux disease,
* Woman pregnant or susceptible to the being,
* Patients deprived of liberty or placed Under the authority of a tutor,
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule,
* Contraindications to the endoscopic procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Suggest that there are significantly more than 60 % of patients with a relative decrease of at least 50 % between the total percentages of esophageal time crossed in pH4 (Ph metric dosage) before and after endoscopic treatment. | 36 months
  Realization of Ph metric dosage (Gastric Ph monitoring)

SECONDARY OUTCOMES:
Rate in percentage of long-term recurrence of high grade dysplasia, low grade dysplasia, or Barrett's oesophagus without dysplasia. | 12 months.
  Realization of several follow-up at 12 months.
Rate in percentage of long-term recurrence of high grade dysplasia, low grade dysplasia, or Barrett's oesophagus without dysplasia. | 24 months.
  Realization of several follow-up at 24 months.
Rate in percentage of long-term recurrence of high grade dysplasia, low grade dysplasia, or Barrett's oesophagus without dysplasia. | 36 months.
  Realization of several follow-up at 36 months.
Evolution of the score of DeMeester of the reflux before and after endoscopic treatment | 36 months.
  Realization of several follow-up from day 1 (post endoscopic resection) to 36 months.
Evolution of the clinical signs of the reflux before and after endoscopic treatment | 36 months.
  Realization of several follow-up from day 1 (post endoscopic resection) to 36 months.
Incidences accumulated of recurrence | 36 months.
  Realization of several follow-up from Day 1 (post endoscopic resection) to 36 months.
Rate of endoscopic complications | 36 months.
  Realization of several follow-up from Day 1 (post endoscopic resection) to 36 months.
Use of Inhibitor of the pump with proton (PPI) | 36 months.
  Realization of several follow-up from Day 1 (post endoscopic resection) to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: CAILLOL Fabrice, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- GENRE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr